CLINICAL TRIAL: NCT02902042
Title: A Randomized Phase I / II Open Label, Multicentre Study of Encorafenib Plus Binimetinib and PD-1 Antibody Pembrolizumab in Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Brief Title: Encorafenib + Binimetinib + Pembrolizumab in Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Acronym: IMMU-TARGET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Dirk Schadendorf (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dirk Schadendorf, Prof. Dr. med., University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-818-201X
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Malignant Melanoma
Keywords: Unresectable or metastatic BRAF V600 mutant melanoma; Encorafenib, binimetinib, pembrolizumab
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Triple therapy (Experimental): Encorafenib, binimetinib and pembrolizumab. Doses as determined in phase I
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Drug: Pembrolizumab
- Arm B: Pembrolizumab alone (Experimental): Pembrolizumab with a dose of 200 mg every 3 weeks.
  Interventions: Drug: Pembrolizumab alone

INTERVENTIONS:
Drug: Encorafenib — Dose determined in phase I. Start dose: 450 mg qd
  Other Names: Braftovi
  Arms: Arm A: Triple therapy
Drug: Binimetinib — Dose determined in phase I. Start dose: 45 mg bid
  Other Names: Mektovi
  Arms: Arm A: Triple therapy
Drug: Pembrolizumab — Dose determined in phase I. Start dose: 200 mg q3w
  Other Names: Keytruda
  Arms: Arm A: Triple therapy
Drug: Pembrolizumab alone — 200 mg q3w
  Other Names: Keytruda
  Arms: Arm B: Pembrolizumab alone

SUMMARY:
This study will investigate the influence of maintenance therapy on progression-free survival (PFS) and overall survival (OS) after combination therapy with BRAF/MEK (MAP-ERK kinase) inhibitors and PD-1 antibody pembrolizumab.

In the safety phase I part the optimal dose of pembrolizumab in combination with BRAF inhibitor and MEK inhibitor and the safety of this three-drugs-combination regime will be determined.

In the randomized part 2 different maintenance therapies will be tested for toxicity and efficacy. Patients with disease control after 6 months of triple therapy will be randomized to receive 2 different maintenance therapies further on, either continuation of triple therapy or administration of pembrolizumab alone.

DETAILED DESCRIPTION:
There is growing interest to understand the best strategies to use targeted therapies and novel immunotherapy for the treatment of advanced melanoma. This study will explore the combination of encorafenib plus binimetinib with the PD-1 antibody pembrolizumab in patients with BRAF mutant melanoma. Combination of two clinically effective approaches, targeting the mutant BRAF pathway by BRAF/MEK inhibition and modulating immunological checkpoint control by administration of a PD-1 antibody, should prolong PFS and OS even further. This study will investigate the influence of maintenance therapy on PFS and OS after triple therapy. Patients with disease control after 6 months of triple therapy will be randomized to receive 2 different maintenance therapies further on to investigate if administration of pembrolizumab only is sufficient for maintenance of disease control. For reasons of safety a phase I study is performed to determine the optimal dosing and schedule of the combination therapy (encorafenib, binimetinib, pembrolizumab).

In the phase II-part, patient will receive triple therapy with the doses defined in phase I for a 6 months induction period. Patients with complete or partial response or stable disease after the 6 months period will be randomized for maintenance therapy:

Arm A: Therapy as in induction period. Arm B: Therapy with pembrolizumab only with a dose of 200 mg every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial.
* Being ≥ 18 years of age on day of signing informed consent.
* Histologically confirmed diagnosis of locally advanced, unresectable or metastatic melanoma AJCC (2017) Stage IIIB, IIIC, IIID or IV with no active brain metastasis. All known CNS lesions must have been only treated with stereotactic therapy or surgery at least 4 weeks prior to the first dose of trial treatment AND they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline); there is no evidence of new or enlarging brain metastases, and the patient must not have used steroids in dosing exceeding 10 mg daily of prednisone equivalent for at least 3 weeks prior to trial treatment.
* Treatment naive patient for locally advanced unresectable or metastatic melanoma. Prior adjuvant or neoadjuvant systemic therapy is permitted (in stage II, III and IV with no evidence of disease) if all related adverse events have either returned to baseline or stabilized.

  (i) Anti-PD-1, anti-CTLA-4, BRAF/MEK inhibitor therapy with at least 6 months between the last dose and date of recurrence.

(ii) Interferon therapy and chemotherapy with the last dose at least 6 weeks prior to registration.

(iii) Radiotherapy with the last radiation at least 28 days prior to registration. Participants must have recovered from all radiation-related toxicities. Note: radiated lesions cannot be used as measurable lesions unless there is clear evidence of progression.

Patients who are in follow-up period of a clinical trial in adjuvant setting may be enrolled.

* Measurable disease, i.e., present with at least one measurable lesion per RECIST, version 1.1, for the definition of a measureable lesion.
* Presence of BRAF mutation V600 in tumor tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion prior to enrollment.
* Performance status of 0 or 1 on the ECOG Performance Scale.
* Adequate organ function: ANC ≥1,500 /mcL, Platelets ≥100,000 / mcL, Hemoglobin ≥9 g/dL OR ≥5.6 mmol/L, Serum creatinine OR Measured or calculated CrCl ≤1.5 X ULN OR ≥50 mL/min for subject with creatinine levels > 1.5 X institutional ULN, Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN, AST and ALT ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases.
* Adequate cardiac function:

  * LVEF ≥ 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram
  * Corrected QT (QTc) interval ≤ 480ms
* All treatment-related toxicities of prior adjuvant or neoadjuvant systemic therapy (except alopecia) must be ≤ Grade 1 according to the CTCAE version 4.03:
* Able to take oral medications.
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use a highly effective form of contraception according to CTFG starting with the first dose of study therapy during the course of this study and for at least 120 days after the last dose of study medication

Exclusion Criteria:

* Currently participating in or having participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Diagnosis of immunodeficiency or receiving systemic steroid therapy in dosing exceeding 10 mg daily of prednisone equivalent or any other form of immunosuppressive therapy within 7 days prior to study Day 1.
* Prior therapy (except if given as adjuvant or neoadjuvant therapy for melanoma) with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways (except for interferon given as adjuvant or neoadjuvant therapy for melanoma).
* Prior therapy (except if given as adjuvant or neoadjuvant therapy for melanoma) with a BRAF inhibitor (including but not limited to vemurafenib, dabrafenib, encorafenib) and / or MEK inhibitor (including but not limited to trametinib, AZD6244, binimetinib, cobimetinib).
* Any previous anti-cancer treatment, extensive radiotherapy or investigational agent for locally advanced unresectable or metastatic melanoma.
* Known additional malignancy that is progressing or required active treatment within 3 years prior to the study.
* Known active CNS metastases and/or carcinomatous meningitis.
* Presence of uveal melanoma.
* History of leptomeningeal metastases.
* History or current evidence of CSR or RVO or predisposing factors to RVO or CSR (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus, history of hyperviscosity or hypercoagulability syndromes).
* History of retinal degenerative disease.
* History of allogeneic bone marrow transplantation or organ transplantation.
* History of Gilbert's syndrome.
* Uncontrolled arterial hypertension despite medical treatment.
* Patients who have neuromuscular disorders associated with elevated creatine kinase (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Impairment of gastrointestinal function or gastrointestinal disease (e.g. ulcerative disease, uncontrolled nausea, vomiting, malabsorption syndrome, small bowel resection).
* Evidence of interstitial lung disease or active, non-infectious pneumonitis or history of (non-infectious) pneumonitis that required steroids.
* Active infection requiring systemic therapy.
* Pregnancy or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit until up to 120 days after the last dose of trial treatment.
* Positive test for HIV.
* Positive test for Hep B or Hep C.
* Receiving a live vaccine within 30 days prior to the first dose of trial treatment.
* Known hypersensitivity reaction to any of the components of study treatment.
* Medical, psychiatric, cognitive or other conditions, including known alcohol or drug abuse that would not permit the subject to complete the study or sign informed consent.
* Patients taking non-topical medication known to be a strong inhibitor of CYP3A4.
* History of life-threatening toxicity related to prior immune therapy (e.g. anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) or kinase inhibition (e.g. BRAF and/or MEK inhibitor) except those that are unlikely to re-occur with standard countermeasures (e.g. hormone replacement after adrenal crisis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of the triple combination treatment] | 42 days
  Dose limiting toxicities (DLT) will be determined within 42 days of therapy start (first pembrolizumab injection) and are defined as all ≥ grade 4 hematological toxicities and certain non-hematological toxicities ≥ CTCAE grade 3.
Phase II: Progression-free survival (PFS) | 24 months
  Time from administration of first study drug to the date of first documented progression (according Recist criteria version 1.1) or death due to any cause, whichever occurs first.
Phase II: PFS rate at 12 months | 12 months
  Rate of patients with PFS after 12 months of therapy
Phase II: PFS rate at 18 months | 18 months
  Rate of patients with PFS after 18 months of therapy
Phase II: PFS rate at 24 months | 24 months
  Number of patients with PFS after 24 months of therapy

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 months
  All adverse events (AEs) / serious adverse events (SAEs) NCI CTCEA (Common Terminology Criteria for Adverse Events) Grade ≥ 3
Objective response rate | 24 months
  Number of patients with complete response (CR), partial response (PR) and stable disease (SD) as best response.
Overall survival time | 24 months
  Time from the date of first administration of study drug to the date of death due to any cause.
1-year survival rate | 12 months
  Number of patients alive in the time period from date of first administration of study drug until 1 year after date of first administration
2-year survival rate | 24 months
  Number of patients alive in the time period from date of first administration of study drug until 2 years after date of first administration

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (11):
- Germany (11):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Augsburg Süd, Augsburg, Bavaria
  - Klinikum rechts der Isar, München, Bavaria
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Universitätsklinikum Gießen und Marburg GmbH, Klinik für Dermatologie und Allergologie, Giessen, Hesse
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - University Hospital Essen, Department of Dermatology, Skin Cancer Center, Essen, North Rhine-Westphalia
  - HELIOS Klinikum Krefeld, Krefeld, North Rhine-Westphalia
  - Gesellschaft für Klinische Forschung Ludwigshafen mbH, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Städtisches Klinikum Dessau, Dessau, Saxony-Anhalt
  - Vivantes Klinikum im Friedrichshain, Friedrichshain, State of Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zimmer L, Livingstone E, Krackhardt A, Schultz ES, Goppner D, Assaf C, Trebing D, Stelter K, Windemuth-Kieselbach C, Ugurel S, Schadendorf D. Encorafenib, binimetinib plus pembrolizumab triplet therapy in patients with advanced BRAFV600 mutant melanoma: safety and tolerability results from the phase I IMMU-TARGET trial. Eur J Cancer. 2021 Nov;158:72-84. doi: 10.1016/j.ejca.2021.09.011. Epub 2021 Oct 13. PMID 34655839